CLINICAL TRIAL: NCT01577147
Title: Generic Protocol for the Collection of Early Pregnancy Urines
Brief Title: Early Pregnancy Sample Collection Study
Acronym: EPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PROTOCOL-0400
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2016-11

CONDITIONS: Pregnancy
Keywords: pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sample collection (Other): Ovulation prediction products provided to aid conception
  Interventions: Other: Ovulation predictions products

INTERVENTIONS:
Other: Ovulation predictions products — Home diagnostics for ovulation prediction will be provided to study volunteers

SUMMARY:
Female volunteers, wishing to become pregnant will be offered the use of Clearblue ovulation prediction products to help identify their most fertile time and aid conception. Volunteers will provide SPD with a daily urine sample throughout the study period, which will be used for the development and validation of SPD products related to pregnancy and fertility.

DETAILED DESCRIPTION:
In order to develop and validate new and existing products SPD needs to maintain a sample bank of early pregnancy urine samples from the beginning of the cycle in which pregnancy is achieved, and throughout pregnancy.

This generic study will be initiated to maintain the SPD sample bank, the study will run continuous to replenish the sample bank, as samples are used.

To obtain these samples, volunteers wishing to become pregnant will be offered the use of a Clearblue ovulation prediction product to enable them to pinpoint their most fertile time and aid conception. Whilst on the study volunteers will be asked to collect daily urine samples and return them to SPD on a regular basis in addition to keeping a daily record of menstrual cycle details and test results. Women who become pregnant during the course of the study will be asked to continue collecting daily urine samples for a minimum of a further 4 weeks. Each volunteer will be on the study for a minimum of 1 and a maximum of 3 cycles. Volunteers will not be allowed to re-enter the study once they have completed without achieving pregnancy

It is anticipated that any one of SPD's marketed ovulation prediction products may be used in this study to aid the conception rate, this may include, but not be limited to the Clearblue fertility monitor and Clearblue digital ovulation test.

It is anticipated SPD will have to recruit approximately 600 volunteers to achieve each 100 pregnancies and that approximately 500 volunteers will be participating at any one time. The study size may be increased or decreased to meet sample demands.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-45
* Have menstrual bleeds
* Seeking to become pregnant
* Willing to provide written, informed consent

Exclusion Criteria:

* Known condition to contra-indicate pregnancy
* Having treatment for infertility.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4025 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Collection of early pregnancy urine samples. | 60 days
  Volunteers who become pregnant during the study will continue to collect daily urine samples until day 60 of the conception cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

REFERENCES:
- [Derived] Gadsby R, Ivanova D, Trevelyan E, Hutton JL, Johnson S. The onset of nausea and vomiting of pregnancy: a prospective cohort study. BMC Pregnancy Childbirth. 2021 Jan 6;21(1):10. doi: 10.1186/s12884-020-03478-7. PMID 33407214
- [Derived] Johnson S, Marriott L, Zinaman M. Can apps and calendar methods predict ovulation with accuracy? Curr Med Res Opin. 2018 Sep;34(9):1587-1594. doi: 10.1080/03007995.2018.1475348. Epub 2018 May 25. PMID 29749274